### **BREATHES:**

# Bringing Respiratory Education for Improved Adherence and Technique Home Through E-Interventions for Self-management

Document date: September 27, 2019

#### **BACKGROUND**

Chronic obstructive pulmonary disease (COPD) results in nearly 750,000 hospitalizations annually and is the third leading cause of 30-day hospital readmissions in the United States. Improving the quality of care for hospitalized COPD patients has recently become a national priority through the Centers for Medicare and Medicaid Services' Hospital Readmissions Reduction Program. A key element of improving care quality is translating existing evidence into improved practice. Extensive evidence exists to support the efficacy of inhaled medications to control and reduce COPD symptoms and to improve patient outcomes. However, the real-world effectiveness of these medications is often limited due both to poor inhaler technique and to insufficient adherence to treatment plans. Not interventions for hospitalized patients with COPD focus on medication reconciliation, treatment optimization, and inhaler technique education prior to being discharged home. However, after discharge home, patients quickly lose inhaler technique skills, have difficulty adhering to complex regimens, and lack tools to aid adherence, such as lung function response to their treatment regimen. Interventions to reinforce skills and support adherence are needed across care transitions to reduce the risk of deleterious health outcomes.

Simple and feasible at-home interventions to provide skills training and adherence support are needed. Our novel idea is to pair at-home inhaler skill training with at-home spirometry measurements to comprehensively support both medication skill and adherence. I propose testing a novel at-home self-management support program called "BREATHES" (Bringing Respiratory Education for improved Adherence and Technique Home through E-interventions for Self-management) Program. BREATHES will include two main components: first, selfdirected inhaler skill training sessions through the virtual Teach-To-Goal (V-TTG) intervention I developed and tested during my K23<sup>32,33</sup> and, second, a handheld lung function device to provide physiologic feedback and capture medication adherence called SpiroPD. 34,35 TTG is a patient-centered strategy that uses cycles of assessment and demonstration tailored to patients' self-management needs; my research shows *in-person* TTG is effective for teaching inhaler technique and reduces acute care utilization. <sup>10,11,18,31,36</sup> *Virtual*-TTG delivers the key features of TTG using virtual patient-directed lessons through novel adaptive technology that provides tailored self-assessment and training. 32,33 My studies demonstrate participants' willingness to use V-TTG at-home for post-discharge booster education and show that V-TTG is effective and may be non-inferior to in-person TTG in significantly reducing inhaler misuse among hospitalized patients. 32-33 However, it remains unknown whether at-home V-TTG sessions will maintain self-management skills over the longer term and how direct physiologic lung monitoring support can impact medication adherence. The proposed studies will determine whether combining at-home skill training with objective measurements of lung function and adherence monitoring through the BREATHES Program improves self-management skills and medication adherence in the first 30 days after hospitalization for COPD.

#### **PURPOSE & HYPOTHESIS**

Our central hypothesis is that patients hospitalized for COPD who subsequently complete the at-home BREATHES Program with V-TTG skill training and SpiroPD adherence support will retain increased medication knowledge, skill, self-efficacy, and adherence that otherwise decays substantially by 30 days post-discharge. To test this hypothesis, I propose the following specific aims:

**SA1.** Determine the feasibility of, adherence to, and efficacy of at-home V-TTG for ongoing inhaler skill training. <u>Hypothesis</u>: Participants who complete both in-hospital and athome V-TTG will have a significantly increased likelihood of demonstrating effective respiratory inhaler technique within 30 days after hospital discharge compared to in-hospital technique.

**SA2.** Determine the feasibility of, adherence to, and efficacy of at-home SpiroPD for COPD medication adherence support. <u>Hypothesis</u>: Participants' use of SpiroPD (PMD Healthcare) will significantly improve their COPD medication adherence.

#### **METHODS OVERVIEW**

We will voluntarily enroll 70 inpatients admitted to the University of Chicago Medicine over the course of 12 months into the at-home BREATHES Program. After obtaining informed consent. participants will complete in-hospital skills, lung function, and medication adherence assessments followed by the BREATHES at-home V-TTG inhaler learning program with selfmonitoring and adherence support through the SpiroPD device. Participants will be trained on V-TTG and SpiroPD use in the hospital. The V-TTG intervention uses novel adaptive learning features that allow learners to participate in tailored educational sessions. They will begin everyother-day lung function assessments using the SpiroPD device in the hospital and continue on discharge. At 48-72 hours after discharge, participants will receive a unique username and password to complete the at-home V-TTG sessions on any of their own desktop or handheld devices; they will complete the V-TTG session at least one time in the first 30 days. Participants will receive reminders for completion of the V-TTG inhaler training and daily lung function monitoring via text messaging Adherence to the at-home V-TTG session (captured through the Smart Sparrow platform), lung function monitoring (captured via the SpiroPD device), and objective inhaler medication adherence (captured via Propeller Health Bluetooth objective monitoring; only 30 of these 70 patients will have objective medication adherence captured) will be assessed throughout the 30-days after discharge via the HIPAA compliant interface. Participants will return at 30 days post-hospital discharge for an in-person evaluation of their inhaler skills, lung function, and acute care utilization.

#### RECRUITMENT

Admission logs (EPIC) at the University of Chicago will be examined each day to screen for potentially eligible inpatients. The treating physician will be contacted for verbal assent using standardized text. Among patients whose physician provides assent, medical records will be reviewed to ascertain eligibility and informed consent will be sought from eligible patients. Approximately 70 patients will be recruited at the University of Chicago Medicine over 12 months.

#### **Study Schema**

| Table 1: Data Collection Tools | | Hospital | Home | 30-day |
|---|---|---|---|---|
| V-TTG adherence | Smart Sparrow platform data capture | _ | Χ | - |
| Inhaler technique | Validated inhaler checklists | Х | - | Χ |
| Inhaler<br>knowledge,<br>efficacy, skills | Inhaler step <i>knowledge</i> , applied inhaler use <i>skill</i> , and <i>attitudes</i> for inhaler self-efficacy assessed through short-answers. | Х | Х | Х |
| Lung function | KoKo® portable spirometer: lung function (FEV1 %predicted). Handheld SpiroPD device (up to daily, at home) | X<br>X | -<br>X | X<br>X |
| Treatment<br>Adherence | Self-reported: Medication adherence report scale (MARS); dose-counter on applicable devices; optional medication diary on the SpiroPD device | Х | - | X |
| 0.16.66 | Objective: Propeller Health® Bluetooth devices. | - | X | X |
| Self-efficacy | "I am confident that I know how to use [inhaler] correctly, (5-point scale). | Х | Х | Х |
| Quality of life (QOL) | The Airway Questionnaire (AQ-20) 20-item tool assesses effect of current symptoms in everyday life for patients with COPD. | Х | - | Х |
| Symptoms | Modified Borg Dyspnea Scale; COPD Severity Score. | Х | - | Χ |
| Health Literacy | Short Test of Functional Health Literacy in Adults: 36 item tool. | Х | - | Χ |

#### **Data Collection Time Points**

- 1. <u>In-Hospital Baseline Assessments.</u> Research Assistant (RA) will assess participants' baseline inhaler technique, inhaler self-efficacy, lung function, and self-reported adherence to their treatment regimen.
- 2. <u>In-Hospital Education:</u> Research Assistant (RA) provides in-person TTG inhaler training and training on how to use the V-TTG and lung function monitoring at home.
- 3. In-Hospital Post-Education Assessments. RA will obtain post-education assessments. 10
- 4. Post-Discharge At-Home BREATHES Program with V-TTG education and lung function monitoring. The participant will complete up to daily lung function (goal of every other day) and medication adherence diaries using the SpiroPD device. The RA will give a unique username and password to each participant to access the V-TTG inhaler training after they have been discharged home. The V-TTG should be completed at least once within the first 30 days after discharge. The RA will send up to three reminders for completion of the lung function monitoring and V-TTG via text messaging. Participants will use their own device (tablet, laptop or desktop computer, or smartphone) for V-TTG use at home. For some patients, data will be collected each time they use their inhaled medication as prescribed. This data will be collected automatically when medication is utilized via a Propeller Health device attached to the inhaler. Patients should use their medication as they are instructed by their provider; no specified usage will be provided by the research team. Only data from regular use will be collected for this portion of the study.
- 5. <u>Post-Discharge Assessments.</u> Thirty days (+/-7 days) after discharge, participants will return for an in-person study visit to assess inhaler technique, adherence measures, lung function, and other assessments.

#### **Device Data Collection**

The SpiroPD device will record participant use and lung function scores. These measurements are stored in a HIPAA compliant server over wifi and are available to the participant and research team. Data from the V-TTG educational modules will be collected via the Smart Sparrow platform. For a subset of approximately 30 patients, a device by Propeller Health will measure objective medication use and adherence. This device will collect only use of an inhaler medication and does not require the participant to use their treatment any differently than prescribed by the clinician. This data will be stored in a HIPPA compliant server only available to the research team.

#### **Survey Data Collection**

Trained research staff will assess the following at the initial enrollment and the 30-day follow-up visit:

- Demographics
- Self-reported treatment adherence
  - MARS
- Self-reported self-efficacy (5-point Likert scale)
- Quality of Life
  - The Airway Questionnaire (AQ-20) 20-item tool assesses effect of current symptoms in everyday life for patients with COPD
- Symptoms
  - Modified Borg Dyspnea Scale

- COPD Severity Tool
- Health Literacy
  - Short Test of Functional Health Literacy in Adults: 36 item tool.

#### **Spirometry**

Spirometry will be performed during the initial visit and during the follow up visit using the portable KoKo spirometer and the SpiroPD device.

#### **DURATION**

Participants will be enrolled in the at-home BREATHES Program for 30 days after discharge from the hospital. They will be in the study for 30 days (with a window of +/- 1 week for the 30 day visit) from the time of enrollment.

#### LOCATION

The study will take place at the University of Chicago Medicine as well as at patient homes.

#### TYPE AND NUMBER OF EXPERIMENTAL SUBJECTS

We will enroll 70 study participants from patients admitted to the University of Chicago Medicine. Only 30 of these 70 subjects will utilize the Propeller Health device to objectively measure medication adherence. This subset of 30 patients will be chosen based on the patients' prescription of a Propeller-compatible inhaler device (as not all inhalers will be compatible with this technology) as well as their willingness to verbally assent to this portion of the study.

#### **Inclusion Criteria**

- 1. Age 18 years and older
- 2. Physician-diagnosed COPD (prior to or during hopsitalization)
- 3. Owns a wifi-enabled device (desktop, laptop, tablet, smartphone, etc.)
- 4. Discharged with a rescue and/or controller MDI
- 5. Visual acuity of at least 20/50 in at least one eye (with or without corrective lens provided by the reseach team for study purposes)

#### **Exclusion Criteria**

- 1. Currently in an intensive care unit
- 2. Physician declines to provide consent
- 3. Patient unable to provide consent (e.g., history of cognitive impairment, unable to understand English) or declines to provide consent

#### STATISTICAL ANALYSES

We will use means, medians, proportions, scatterplots, and histograms to describe the data. We will test for group differences using the *t*-test, the Wilcoxon rank sum test, Pearson's chi-squared test, or Fisher's exact tests, as appropriate. The primary outcomes for Aim 1 are athome V-TTG adherence and inhaler technique and for Aim 2, at-home lung function testing adherence and medication adherence. McNemar's chi-squared tests will be used to compare 30 day post-discharge vs. pre-discharge adherence to the devices, prevalence of inhaler misuse (≤10/12 steps correct), and medication adherence. Secondary outcomes will include change in

self-efficacy for inhalers, symptom burden, self-reported utilization of health care services, and QOL. A two-tailed p-value less than 0.05 will define statistical significance.

#### POTENTIAL RISKS AND BENEFITS

The subject may be uncomfortable answering some interview questions. All subjects will be told that they can refuse to answer any question.

Loss of confidentiality. To help ensure that patients' health information remains private, we will restrict access to data collected for our study to study personnel only (via use of password-protection and locked cabinets for study documents). Study ID numbers will be generated and will be used when discussing and/or reviewing data at study meetings. Also, study reports will report results in aggregate and not contain information that can be used to identify individual patients.

Spirometry is safe and is commonly used to measure disease severity but can cause some minor chest soreness or lightheadedness.

#### **DATA SAFETY MONITORING PLAN**

A Data and Safety Monitoring Board will be formed to protect the safety of study subjects to ensure that they are not exposed to undue risk and to assure that the quality of the research data generated is acceptable and protected. The DSMB will operate without any conflicts of interest and/or undue influence from interested parties including the study investigators and funder. The DSMB members' primary responsibilities will be to ensure sufficient progress and implementation of the project and to ensure safety of the participants. This work will include evaluations of patient accrual rates during the recruitment period, patient safety including adverse and/or unplanned events, and the integrity of the data collection and management during this study. All serious adverse events will be forwarded to the IRB and DSMB within 48 hours of being recognized by study staff. The DSMB will have authority to recommend modifications to the clinical investigations or to stop these investigations if there are concerns with patient safety or the integrity of the study.

Study investigators will communicate with the DSMB members about the study only as needed to make decisions related to meetings and meeting materials. Communication between DSMB members will be initiated by the DSMB chair. Communication with NHLBI will led by the DSMB chair and/or PI depending on the circumstances of the required communication such as communication regarding the DSMB report. This DSMB will consist of 3 members, including two faculty at the University of Chicago and one from Northwestern, who will be involved with the safety and monitoring of this study: Kenzie Cameron, PhD, Peter O'Donnell MD, and Matthew Churpek MD. PhD. All board members will meet our institution's requirements for declaring conflicts of interest. The DSMB will convene initially to review, provide feedback on, and ultimately approve the data safety monitoring plan prior to beginning enrollment. The board will then meet half way through the enrollment period or when we reach 50% enrollment, whichever comes first. The NHLBI Program Office will be notified of scheduled meeting in advance should the program manager and/or delegate wish to monitor the meeting. A report of these minutes will be forwarded to the PI and to NIH NHLBI staff. A summary of DSMB deliberations and recommendations will be submitted to the IRB. Additional DSMB meetings may be scheduled as needed.

## POTENTIAL BENEFITS OF THE PROPOSED RESEARCH TO THE PARTICIPANTS AND OTHERS

Although we do not believe that participants will directly benefit from this study, beyond potential improved aderence, self-monitoring, and inhaler technique skills, the risks are reasonable in

relation to the benefits because the proposed studies could help us learn about better ways to patients to self-assess their lung function and continue to learn self-management skills after they transition home post-discharge.

#### CONFIDENTIALITY

We understand the importance of protecting the confidentiality of information from our research participants. We will use unique alphanumeric identifiers for the data collection process. These unique codes will link all related participant information. All case report forms will be stored in locked file cabinets. All electronic data will be secured using password-protected files. Access to these data will be restricted to the research staff only. Analytic files will not contain any identifying information. All reports/manuscripts will be prepared in such a way that individual patients will not be identifiable. Additional specific details are described above.

#### **COMPENSATION**

Participants will receive compensation for their time (\$25 inpatient, \$50 30-day in-person visit).

Additionally, study participants will receive the SpiroPD for use during the study and will be able to keep this device for their personal use upon completion of the study; this device is valued at \$500.

#### **INFORMED CONSENT**

Medical records at the University of Chicago will be examined each day to screen for potentially eligible patients. The treating physician will be contacted for verbal or written assent using standardized text. To reduce the burden on busy clinicians of individual pages/phone calls for assent, we will also provide additional options for assent ahead of clinical rotations (see X). Among patients whose physician provides assent, medical records will be reviewed to ascertain eligibility and written informed consent will be sought from eligible patients.

#### **REFERENCES**

- National Center for Health Statistics. Chronic Obstructive Pulmonary Disease (COPD) Includes: Chronic Bronchitis and Emphysema. http://www.cdc.gov/nchs/fastats/copd.htm. Last updated May 3, 2017 Accessed February 6, 2018.
- Jencks SF, Williams MV, Coleman EA. Rehospitalizations Among Patients in the Medicare Fee-for-Service Program. N Engl J Med. 2009;360(14):1418-1428.
- Centers for Medicare and Medicaid Services. Hospital Readmissions Reduction Program. https://www.cms.gov/medicare/medicare-fee-for-service-payment/acuteinpatientpps/readmissions-reduction-program.html. Published April 18, 2016. Accessed March 12, 2017.
- Feemster LC, Au DH. Penalizing hospitals for chronic obstructive pulmonary disease readmissions. Am J Respir Crit Care Med. 2014;189(6):634-639.
- Wagner EH, Austin BT, Davis C, Hindmarsh M, Schaefer J, Bonomi A. Improving chronic illness care: translating evidence into action. Health Aff Proj Hope. 2001;20(6):64-78.
- 6. Avorn J, Fischer M. "Bench to behavior": translating comparative effectiveness research into improved clinical practice. *Health Aff Proj Hope*. 2010;29(10):1891-1900.
- 7. Rand CS. Patient adherence with COPD therapy. Eur Respir Rev. 2005;14(96):97-101.
- 8. George J, Kong DCM, Stewart K. Adherence to disease management programs in patients with COPD. *Int J Chron Obstruct Pulmon Dis.* 2007;2(3):253-262.
- 9. Zwerink M, Brusse-Keizer M, van der Valk PD, Zielhuis GA, Monninkhof EM, van der Palen J, Frith PA, Effing T. Self management for patients with chronic obstructive pulmonary disease. *Cochrane Database Syst Rev.* 2014;(3):CD002990.
- Press VG, Arora VM, Shah LM, Lewis SL, Charbeneau J, Naureckas ET, Krishnan JA. Teaching the use of respiratory inhalers to hospitalized patients with asthma or COPD: a randomized trial. *J Gen Intern Med*. 2012;27(10):1317-1325.
- Press VG, Arora VM, Trela KC, Adhikari R, Zadravecz FJ, Liao C, Naureckas E, White SR, Meltzer DO, Krishnan JA. Effectiveness of Interventions to Teach Metered-Dose and Diskus Inhaler Techniques. A Randomized Trial. *Ann Am Thorac Soc.* 2016;13(6):816-824.

- 12. Bourbeau J, Julien M, Maltais F, Rouleau M, Beaupré A, Bégin R, Renzi P, Nault D, Borycki E, Schwartzman K, Singh R, Collet JP; Chronic Obstructive Pulmonary Disease axis of the Respiratory Network Fonds de la Recherche en Santé du Québec. Reduction of hospital utilization in patients with chronic obstructive pulmonary disease: a disease-specific self-management intervention. *Arch Intern Med.* 2003;163(5):585-591.
- Gadoury MA, Schwartzman K, Rouleau M, Maltais F, Julien M, Beaupré A, Renzi P, Bégin R, Nault D, Bourbeau J;
   Chronic Obstructive Pulmonary Disease axis of the Respiratory Health Network, Fonds de la recherche en santé du Québec (FRSQ). Self-management reduces both short- and long-term hospitalisation in COPD. Eur Respir J. 2005:26(5):853-857.
- 14. GOLD 2017 Global Strategy for the Diagnosis, Management and Prevention of COPD. http://goldcopd.org/gold-2017-global-strategy-diagnosis-management-prevention-copd/. Accessed March 12, 2017.
- Hanania NA, Darken P, Horstman D, Reisner C, Lee B, Davis S, Shah T. The efficacy and safety of fluticasone propionate (250 microg)/salmeterol (50 microg) combined in the Diskus inhaler for the treatment of COPD. *Chest.* 2003;124(3):834-843
- 16. Celli BR, Thomas NE, Anderson JA, Ferguson GT, Jenkins CR, Jones PW, Vestbo J, Knobil K, Yates JC, Calverley PM. Effect of pharmacotherapy on rate of decline of lung function in chronic obstructive pulmonary disease: results from the TORCH study. Am J Respir Crit Care Med. 2008;178(4):332-338.
- 17. Lavorini F, Magnan A, Dubus JC, Voshaar T, Corbetta L, Broeders M, Dekhuijzen R, Sanchis J, Viejo JL, Barnes P, Corrigan C, Levy M, Crompton GK. Effect of incorrect use of dry powder inhalers on management of patients with asthma and COPD. *Respir Med.* 2008;102(4):593-604.
- 18. Press VG, Arora VM, Shah LM, Lewis SL, Ivy K, Charbeneau J, Badlani S, Nareckas E, Mazurek A, Krishnan JA. Misuse of respiratory inhalers in hospitalized patients with asthma or COPD. *J Gen Intern Med.* 2011;26(6):635-642.
- Roggeri A, Micheletto C, Roggeri DP. Inhalation errors due to device switch in patients with chronic obstructive pulmonary disease and asthma: critical health and economic issues. *Int J Chron Obstruct Pulmon Dis.* 2016;11:597-602.
- Vanderman AJ, Moss JM, Bailey JC, Melnyk SD, Brown JN. Inhaler misuse in an older adult population. Consult Pharm J Am Soc Consult Pharm. 2015;30(2):92-100.
- 21. Bonds RS, Asawa A, Ghazi Al. Misuse of medical devices: a persistent problem in self-management of asthma and allergic disease. *Ann Allergy Asthma Immunol*. 2015 Jan;114(1):74-76.e2.
- 22. Batterink J, Dahri K, Aulakh A, Rempel C. Evaluation of the use of inhaled medications by hospital inpatients with chronic obstructive pulmonary disease. *Can J Hosp Pharm.* 2012;65(2):111-118.
- 23. Melani AS, Canessa P, Coloretti I, DeAngelis G, DeTullio R, Del Donno M, Giacobbe R, Scarlato I, Serafini A, Barbato N, Vaghi A, Sestini P; Educational Study Group of the Italian Association of Hospital Pulmonologists (AIPO). Inhaler mishandling is very common in patients with chronic airflow obstruction and long-term home nebuliser use. *Respir Med*. 2012;106(5):668-676.
- 24. Melani AS, Bonavia M, Cilenti V, Cinti C, Lodi M, Martucci P, Serra M, Scichilone N, Sestini P, Aliani M, Neri M; Gruppo Educazionale Associazione Italiana Pneumologi Ospedalieri. Inhaler mishandling remains common in real life and is associated with reduced disease control. *Respir Med.* 2011;105(6):930-938.
- 25. Melani AS1, Zanchetta D, Barbato N, Sestini P, Cinti C, Canessa PA, Aiolfi S, Neri M; Associazione Italiana Pneumologi Ospedalieri Educational Group. Inhalation technique and variables associated with misuse of conventional metered-dose inhalers and newer dry powder inhalers in experienced adults. *Ann Allergy Asthma Immunol.* 2004;93(5):439-46.
- McFadden ER. Improper patient techniques with metered dose inhalers: clinical consequences and solutions to misuse. J Allergy Clin Immunol. 1995;96(2):278-283.
- 27. Bhatt SP, Wells JM, Iyer AS, Kirkpatrick DP, Parekh TM, Leach LT, Anderson EM, Sanders JG, Nichols JK, Blackburn CC, Dransfield MT. Results of a Medicare Bundled Payments for Care Improvement Initiative for COPD Readmissions. *Ann Am Thorac Soc.* 2017;14(5):643-648.
- Zafar MA, Panos RJ, Ko J, Otten LC, Gentene A, Guido M, Clark K, Lee C, Robertson J, Alessandrini EA. Reliable adherence to a COPD care bundle mitigates system-level failures and reduces COPD readmissions: a system redesign using improvement science. BMJ Qual Saf. 2017;26(11):908-918.
- 29. Parikh R, Shah TG, Tandon R. COPD exacerbation care bundle improves standard of care, length of stay, and readmission rates. *Int J Chron Obstruct Pulmon Dis.* 2016;11:577-583.
- 30. George J, Kong DCM, Thoman R, Stewart K. Factors associated with medication nonadherence in patients with COPD. *Chest.* 2005;128(5):3198-3204.
- 31. Paasche-Orlow MK, Riekert KA, Bilderback A, Chanmugam A, Hill P, Rand CS, Brancati FL, Krishnan JA. Tailored Education May Reduce Health Literacy Disparities in Asthma Self-Management. *Am J Respir Crit Care Med*. 2005;172(8):980-986.
- 32. Press VG, Kelly CA, Kim JJ, White SR, Meltzer DO, Arora VM. Virtual Teach-To-Goal<sup>™</sup> Adaptive Learning of Inhaler Technique for Inpatients with Asthma or COPD. *J Allergy Clin Immunol Pract*. 2017;5(4):1032-1039.e1.
- Wu M, Woodrick N, Arora VM, Farnan JM, Press VG. Developing a Virtual Teach-To-Goal Inhaler Technique Learning Module: A Mixed Methods Approach. J Allergy Clin Immunol Pract. 2017;5(6):1728-1736. J
- 34. Shakkottai A, Nasr SZ. The Use of Home Spirometry in Pediatric Cystic Fibrosis Patients: Results of a Feasibility Study. *Glob Pediatr Health*. 2017;4:2333794X17690315.
- 35. Henriques C. Children with Cystic Fibrosis Who Use Spiro PD at Home Improve Lung Function, Study Shows. Cystic Fibrosis News Today. https://cysticfibrosisnewstoday.com/2017/04/25/home-use-of-spiro-pd-improves-lung-function-of-children-with-cystic-fibrosis/. April 2017. Accessed October 4, 2017.
- Kripalani S, Bengtzen R, Henderson LE, Jacobson TA. Clinical research in low-literacy populations: using teach-back to assess comprehension of informed consent and privacy information. *IRB*. 2008;30(2):13-19.